CLINICAL TRIAL: NCT00132834
Title: Exhaled Breath Condensates ("EBC") Study: Research Plan NIH/NIAID: Inner City Asthma Consortium (ICAC)
Brief Title: Methods of Determining Asthma Severity in Children
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT ICAC-05
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Asthma/no ICS: Asthmatic children who are not currently taking ICS
  Interventions: Device: R-Tube or EcoScreen
- Asthma/ICS: Asthmatic children on ICS
  Interventions: Device: R-Tube or EcoScreen
- Non-asthmatic children: Children without asthma
  Interventions: Device: R-Tube or EcoScreen

INTERVENTIONS:
Device: R-Tube or EcoScreen — Device for collection of exhaled breath condensates (EBC) collection (i.e. condensing and collecting breath vapor from a cold, solid surface)

SUMMARY:
Current methods of measuring asthma severity can be problematic when used with children. A measurement called exhaled breath condensates (EBC) may be a more useful way to determine asthma severity in childhood. The purpose of this study is to determine if EBC measurements are useful for determining asthma severity in asthmatic children as compared to currently used laboratory measures.

Study hypotheses: 1) A broad panel of EBC measures will distinguish asthmatic children not on inhaled corticosteroids (ICS) from both asthmatic children routinely taking ICS and nonasthmatic controls. 2) Standardized equipment and methodologies for EBC collection, processing, storage, shipping, and pH and mediator measurements can be developed that will eliminate significant contamination from oropharyngeal saliva and allow for shipping and processing at a central site.

DETAILED DESCRIPTION:
The current national guidelines for assessing asthma severity have several limitations for use in asthmatic children. One major limitation is that spirometric measures of airflow limitation, including forced expiratory volume in one second (FEV1), generally cannot be reliably obtained in children less than 7 years of age. Furthermore, most children with asthma have essentially normal measures of airflow by spirometry or peak flow, so such measurements are generally not useful in diagnosis and treatment. Previous studies indicate that lung-specific biomarkers of inflammation, such as bronchial hyperresponsiveness measures, might simplify, improve, and optimize the guidelines. Collection of EBC samples may also be useful; EBC samples can be obtained by noninvasive means and are easier to obtain than conventional samples. However, contamination by saliva is an issue in collecting EBC samples, and standardization of sample collection is needed. This study will compare the utility of two different sample collecting equipment, the EcoScreen and the R-Tube. This study will also evaluate the usefulness of EBC samples in distinguishing between asthmatic children taking ICS, asthmatic children not taking ICS, and nonasthmatic children.

There are 2 parts to this study. In Part A, two EBC samples will be collected from each participant. Some participants will be have one EBC sample taken by the EcoScreen and the other taken by the R-Tube; other participants will have both samples taken by the R-Tube. In Part B, asthmatics taking ICS, asthmatics not taking ICS, and nonasthmatics will give 2 EBC samples each via the R-Tube.

Participants will be asked to complete a questionnaire on their asthma symptoms and allergies and will have a brief physical exam. Allergy skin prick testing, urine collection, measurement of exhaled nitric oxide, and conventional incentive spirometry (used to obtain several measures of lung function) will also occur. Participants will also be asked to donate a blood sample.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Physician-diagnosed asthma
* Symptoms consistent with persistent asthma in the year prior to study entry
* Able to speak and understand English
* Parent or guardian willing to provide informed consent

Exclusion Criteria for All Participants:

* Diagnoses indicating other lung-related disorders (e.g., cystic fibrosis, bronchopulmonary dysplasia [BPD])
* Allergy to latex
* Smoker
* Albuterol use within 12 hours of study entry
* Long-acting bronchodilator or leukotriene modifier use within 24 hours of study entry
* Unable to use the R-Tube. More information on this criterion can be found in the DAIT ICAC-EBC protocol.

Exclusion Criteria for Part A Participants:

* ICS or oral corticosteroid use in the month prior to study entry

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2003-11; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H. Liu, MD, Principal Investigator — National Jewish Health; Wayne Morgan, MD, CM, Principal Investigator — University of Arizona Health Sciences Center

REFERENCES:
- [Background] Baraldi E, Ghiro L, Piovan V, Carraro S, Zacchello F, Zanconato S. Safety and success of exhaled breath condensate collection in asthma. Arch Dis Child. 2003 Apr;88(4):358-60. doi: 10.1136/adc.88.4.358. PMID 12651772
- [Background] Covar RA, Szefler SJ, Martin RJ, Sundstrom DA, Silkoff PE, Murphy J, Young DA, Spahn JD. Relations between exhaled nitric oxide and measures of disease activity among children with mild-to-moderate asthma. J Pediatr. 2003 May;142(5):469-75. doi: 10.1067/mpd.2003.187. PMID 12756375
- [Background] Szefler SJ, Apter A. Advances in pediatric and adult asthma. J Allergy Clin Immunol. 2005 Mar;115(3):470-7. doi: 10.1016/j.jaci.2004.12.1123. PMID 15753890